CLINICAL TRIAL: NCT01775306
Title: Not Invasive Monitoring at Cardiac Recompensation
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 10-081
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Cardiac Recompensation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to find out if data can be provided by external sensor technology which is suitable for controlling the therapy of patients with cardiac recompensation.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute or chronic cardiac decompensation with and without pulmonary oedema
* male and female patients aged at least 18 years

Exclusion Criteria:

* pregnancy or breast feeding
* implanted pacemaker / CRT / ICD exept Medtronic OptiVol
* patients being unable to consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiac recompensation
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
suitable Data | 15 minutes per day and per patient, 3-5 days, at most 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy Hospital Aachen, Aachen, North Rhine Westfalia, Germany